CLINICAL TRIAL: NCT01818492
Title: A Phase 2/3 Open-label Single Arm Multicentre Study to Assess Safety Tolerability Pharmacokinetics and Efficacy of i.v. Administrations of NI-0501 an Anti-IFNγ mAb in Paediatric Patients With Primary Haemophagocytic Lymphohistiocytosis
Brief Title: Study to Investigate Safety, Efficacy of an Anti-IFNγ mAb in Children With Primary Haemophagocytic Lymphohistiocytosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Seventh Framework Programme (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI-0501-04; 2012-003632-23 (EudraCT Number)
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2021-04

CONDITIONS: Primary Haemophagocytic Lymphohistiocytosis
Keywords: Emapalumab
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Emapalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NI-0501 (Experimental): NI-0501 administered by IV infusion at a starting dose of 1 mg/kg.
  Interventions: Biological: NI-0501

INTERVENTIONS:
Biological: NI-0501

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of a new drug aimed at controlling disease activity in patients diagnosed with primary haemophagocytic lymphohistiocytosis. The new drug can be administered as the first-line therapy, to patients not previously treated with the current standard of care, or can be given to patients who have either failed or were unable to tolerate the current standard of care. Administration will be on top of a glucocorticosteroid, which is usually part of the current recommended treatment.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, tolerability and efficacy of a new drug aimed at controlling disease activity in patients diagnosed with primary haemophagocytic lymphohistiocytosis. The new drug can be administered as the first-line therapy, to patients not previously treated with the current standard of care, or can be given to patients who have either failed or were unable to tolerate the current standard of care. Administration will be on top of a glucocorticosteroid, which is usually part of the current recommended treatment.

All participants in the NI-0501-04 study (NCT01818492) were invited to participate in the long-term follow-up study NI-0501-05 (NCT02069899). For the primary completion date, mentioned here, we refer to the NI-0501-04 study, even though in accordance with the NI-0501-04 study objectives, namely the assessment of long-term efficacy and safety endpoints, the study analyses also included data collected in the long-term follow-up study NI-0501-05. Hence these data are reported together. Study NI-0501-05 accepts patients from NI-0501-04 and NI-0501-06. Data collection for the patients from NI-0501-04 is completed.

The primary efficacy and safety analyses are based on the regulatory cut-off date of 20 July 2017. Refer to the publication in N Engl J Med 2020 May 7; 382 (19):1811-1822. Follow-on analyses have been conducted on all patients enrolled in the study, i.e. including the patients enrolled after the cut-off date of 20 July 2017. The results reported here refer to the totality of the 45 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male and female
* Age: up to and including 18 years at diagnosis of Haemophagocytic Lymphohistiocytosis
* Primary HLH patients
* Patient (if ≥ 18 years old), or patient's legal representative(s) must have signed informed consent

Exclusion Criteria:

* Diagnosis of secondary Haemophagocytic Lymphohistiocytosis consequent to a proven rheumatic or neoplastic disease.
* Body weight < 3 kg.
* Patients treated with biologics within a specific timeframe
* Active Mycobacteria, Histoplasma Capsulatum, Shigella, Salmonella, Campylobacter and Leishmania infections.
* Presence of malignancy.
* Concomitant disease or malformation severely affecting the cardiovascular, pulmonary, liver or renal function

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Radmila Kanceva, MD, Study Director — Swedish Orphan Biovitrum
Locations (20):
- United States (8):
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I. duPont Hospital for Children - Nemours Center for Cancer and Blood Disorders - Division of Pediatric Hematology Oncology, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital - Division of Immunobiology - Department of Pediatrics, Cincinnati, Ohio
  - Texas Children's Cancer Center, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- University Children's Hospital, Münster, Germany
- Italy (6):
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - Istituto Giannina Gaslini, Genoa
  - Azienda Ospedaliera San Gerardo, Monza
  - Azienda Ospedaliera Padova - Clinica di Oncoematologia Pediatrica, Padua
  - Ospedale Pediatrico Bambino Gesu', Roma
  - Ospedale Donna Bambino - U.O.C. Oncoematologia Pediatrica, Verona
- Spain (3):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Niño Jesús, Madrid
- Karolinska University Hospital, Stockholm, Sweden
- Great Ormond Street Hospital - Department of Haematology, London, United Kingdom

REFERENCES:
- [Derived] Brossard P, Laveille C. Population Pharmacokinetics of the Anti-Interferon-Gamma Monoclonal Antibody Emapalumab: An Updated Analysis. Rheumatol Ther. 2024 Jun;11(3):869-880. doi: 10.1007/s40744-024-00669-y. Epub 2024 Apr 25. PMID 38662147
- [Derived] Locatelli F, Jordan MB, Allen C, Cesaro S, Rizzari C, Rao A, Degar B, Garrington TP, Sevilla J, Putti MC, Fagioli F, Ahlmann M, Dapena Diaz JL, Henry M, De Benedetti F, Grom A, Lapeyre G, Jacqmin P, Ballabio M, de Min C. Emapalumab in Children with Primary Hemophagocytic Lymphohistiocytosis. N Engl J Med. 2020 May 7;382(19):1811-1822. doi: 10.1056/NEJMoa1911326. PMID 32374962
- See also: NI-0501-05, long-term follow-up study description on clinicaltrials.gov — https://www.clinicaltrials.gov/ct2/show/NCT02069899

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were screened within 1 week prior to the first administration of emapalumab (NI-0501). 66 patients were screened, and 45 were enrolled and treated.
Groups:
- NI-0501: All patients received emapalumab at a starting dose of 1 mg/kg every 3 days with possible escalation up to 10 mg/kg, for a minimum of 4 weeks.
Period: Overall Study
Arm/Group | NI-0501
Started | 45
Completed | 35
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1
Not completed — Additional therapy when not allowed PP | 4

BASELINE CHARACTERISTICS:
Arm/Group | NI-0501
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 1 [0.1 to 13]
Age, Customized [Count of Participants; unit: Participants]
  <2 years | 32
  ≥ 2 - < 12 years | 12
  ≥ 12 - <18 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30
  Asian | 7
  African Descent | 3
  Mixed/multi-racial | 0
  LOther | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23
  Europe | 22
HLH disease chracteristics at baseline [Count of Participants; unit: Participants]
  Fever | 6
  Splenomegaly | 27
  Platelet counts < 100 x10^9/L | 31
  Neutrophil counts < 1 x10^9/L | 25
  Ferritin > 500 μg/L | 38
  Ferritin > 2000 μg/L | 30
  Fibrinogen < 1.5 g/L | 20
  Triglycerides > 3 mmol/L | 29
  D-Dimers > 500 μg/L | 33
  ALT > 125 IU/L | 21
  Total bilirubin > 25 μmol/L | 13
  LDH > 1000 IU/L | 12
  CNS involvement | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Second Line
Description: Achievement of either Complete (CR) or Partial Response (PR), or HLH Improvement (HI) at End of Treatment of Study NI 0501-04 (EOT 04), based on pre-specified algorithm.
  CR: no fever, normal spleen size, no cytopenia (ANC ≥ 1.0x109/L and platelet count ≥ 100x109/L), no hyperferritinemia (serum ferritin <2000 μg), no coagulopathy (normal D-dimer and/or fibrinogen >150 mg/dL), no neurological and CSF abnormalities attributed to HLH, no sustained worsening of sCD25.
  PR: at least 3 HLH clinical and laboratory criteria (including CNS abnormalities) met the CR criteria, no progression of other aspects of HLH disease pathology.
  HI: improvement (>50% change from baseline) of at least 3 HLH clinical and laboratory criteria (including CNS involvement).
Time Frame: End of Treatment (3 days after the last infusion of emapalumab in study NI-0501-04, occurring between 4 and 8 weeks)
Population: Primary analysis set: Second Line (27 patients who had previously received conventional HLH therapy before enrollment, data collected by regulatory cut-off: 20 July 2017)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NI-0501
Number analyzed (Participants) | 27
percentage of participants | 63.0 [42.4 to 80.6]
Statistical Analysis 1: Comparison: NI-0501; Pre-specified null hypothesis that ORR is at most 40%; Test type: Superiority; p = 0.0134, Exact binomial test; This test was undertaken at the one-sided 0.025 significance level

2. Primary Outcome: Overall Response Rate (ORR) All Treated
Description: as for outcome 1
Time Frame: End of Treatment (3 days after the last infusion of emapalumab in study NI-0501-04, occurring between 4 and 8 weeks)
Population: Primary analysis set: All Treated (all patients who received any part of an emapalumab infusion, data collected by regulatory cut-off: 20 July 2017)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NI-0501
Number analyzed (Participants) | 34
percentage of participants | 64.7 [46.5 to 80.3]
Statistical Analysis 1: Comparison: NI-0501; Pre-specified null hypothesis that ORR is at most 40%; Test type: Superiority; p = 0.0031, Exact binomial test; This test was undertaken at the one-sided 0.025 significance level

3. Primary Outcome: Overall Response Rate (ORR) Follow-on Analysis Set:
Description: as for outcome 1
Time Frame: End of Treatment (3 days after the last infusion of emapalumab in study NI-0501-04, occurring between 4 and 8 weeks)
Population: Follow-on analysis set: Second Line (34 patients who had previously received conventional HLH therapy before enrollment, totality of the data collected in the NI-0501-04 study)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NI-0501
Number analyzed (Participants) | 34
percentage of participants | 58.8 [40.7 to 75.4]
Statistical Analysis 1: Comparison: NI-0501; Pre-specified null hypothesis that ORR is at most 40%; Test type: Superiority; p = 0.0205, Exact binomial test; This test was undertaken at the one-sided 0.025 significance level

4. Primary Outcome: Overall Response Rate (ORR) at End of Treatment in Study NI-0501-04 (EOT 04) Follow-on Analysis Set: All Treated
Description: as for outcome 1
Time Frame: End of Treatment (3 days after the last infusion of emapalumab in study NI-0501-04, occurring between 4 and 8 weeks)
Population: Follow-on analysis set: All Treated (45 patients who received any part of an emapalumab infusion, totality of the data collected in the NI-0501-04)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NI-0501
Number analyzed (Participants) | 45
percentage of participants | 60.0 [44.3 to 74.3]
Statistical Analysis 1: Comparison: NI-0501; Pre-specified null hypothesis that ORR is at most 40%; Test type: Superiority; p = 0.0053, Exact binomial test; This test was undertaken at the one-sided 0.025 significance level

5. Secondary Outcome: Time to Response
Description: Time from the date of the first dose of emapalumab to first achievement of response (at least HLH improvement)
Time Frame: Assessed up to End of Treatment (3 days after the last infusion of emapalumab in study NI-0501-04, occurring between 4 and 8 weeks)
Population: All Treated (all patients who received any part of an emapalumab infusion)
Measure: Median (95% Confidence Interval); unit: Count of days
Arm/Group | NI-0501
Number analyzed (Participants) | 45
Count of days | 7.0 [6.0 to 9.0]

6. Secondary Outcome: Durability of First Response
Description: Maintenance of response achieved any time during the study
Time Frame: as for outcome 5
Population: All Treated (all patients who received any part of an emapalumab infusion)
Measure: Median (95% Confidence Interval); unit: Count of days
Arm/Group | NI-0501
Number analyzed (Participants) | 45
Count of days | 58.0 [39.0 to NA] — Upper limit of 95% CI is not estimable due to too few events.

7. Secondary Outcome: Overall Survival
Description: Number of patients being alive at end of treatment or at week 8, pending on which comes first.
Time Frame: Time from the date of first dose to last dose, or 8 weeks after first dose.
Population: All Treated (all patients who received any part of an emapalumab infusion)
Measure: Number; unit: participants
Arm/Group | NI-0501
Number analyzed (Participants) | 45
participants | 42

8. Secondary Outcome: Number of Patients Able to Reduce Glucocorticoids
Description: Number of patients able to reduce glucocorticoids by 50% or more and between ≥30%-<50%, of baseline dose at EOT 04.
Time Frame: End of Treatment (3 days after the last infusion of emapalumab in study NI-0501-04, occurring between 4 and 8 weeks.
Population: All Treated (all patients who received any part of an emapalumab infusion)
Measure: Number; unit: Percentage of patients
Arm/Group | NI-0501
Number analyzed (Participants) | 45
Percentage of patients
  Reduction ≥50% | 46.7
  Reduction ≥30%-<50% | 11.1

9. Secondary Outcome: Cumulative Duration of Response
Description: Percent of treatment time in response from the first achievement of an Overall Response until HSCT conditioning, or End of Treatment 04/05 (if the patient did not have HSCT performed) Where applicable, data were collected in both NI-0501-04 and long-term follow-up study NI-0501-05.
Time Frame: up to start of HSCT conditioning, whenever HSCT conditioning is scheduled (at least 4 weeks after treatment start), or End of Treatment 04/05 (if the patient did not have HSCT performed)
Population: All Treated (all patients who received any part of an emapalumab infusion)
Measure: Median (Inter-Quartile Range); unit: Percentage of treatment time
Arm/Group | NI-0501
Number analyzed (Participants) | 45
Percentage of treatment time | 78.6 [33.3 to 91.9]

10. Secondary Outcome: Survival Pre-HSCT
Description: Time from the date of first dose to the date of death, expressed in Kaplan-Meier survival probability estimates. Patients who receive HSCT will be censored at that date; patients who did not receive HSCT will be censored at last date of contact.
  Where applicable, data were collected in both NI-0501-04 and long-term follow-up study NI-0501-05.
Time Frame: Assessed up to HSCT, whenever HSCT occurred (up to approximately 6 months after treatment initiation)
Population: All Treated (all patients who received any part of an emapalumab infusion)
Measure: Number (95% Confidence Interval); unit: Kaplan-Meier survival probability
Arm/Group | NI-0501
Number analyzed (Participants) | 45
Kaplan-Meier survival probability
  Month 3: number analyzed (Participants) | 35
  Month 3 | 0.83 [0.669 to 0.915]
  Month 6: number analyzed (Participants) | 35
  Month 6 | 0.73 [0.524 to 0.859]

11. Secondary Outcome: Survival Post-HSCT
Description: Time from the date of first dose to the date of death, expressed in Kaplan-Meier survival probability estimates. Patients without an event will be censored at last assessment date in either the NI-0501-04 or NI-0501-05 study. Patients who do not proceed to HSCT will be excluded from this analysis.
Time Frame: Assessed up to Last Observation (up to 1 year after transplant, or up to approximately 18 months after treatment initiation)
Population: All Treated (all patients who received any part of an emapalumab infusion)
Measure: Number (95% Confidence Interval); unit: Kaplan-Meier survival probability
Arm/Group | NI-0501
Number analyzed (Participants) | 45
Kaplan-Meier survival probability
  Month 6: number analyzed (Participants) | 24
  Month 6 | 0.82 [0.621 to 0.921]
  Month 12: number analyzed (Participants) | 24
  Month 12 | 0.82 [0.621 to 0.921]

ADVERSE EVENTS:
Time Frame: Assessed up to Last Observation (up to 1 year after HSCT, or up to approximately 18 months after treatment initiation).
Description: Adverse Events are summarized for the NI-0501-04 and long-term follow-up NI-0501-05 studies, and analyzed separately for the pre-conditioning and post-conditioning time periods .
Groups:
- Pre-conditioning: All patients before start of conditioning. Conditioning is the treatments used to prepare a patient for stem cell transplantation.
- Post-conditioning: All patients after start of conditioning. Conditioning is the treatments used to prepare a patient for stem cell transplantation.
Arm/Group | Pre-conditioning | Post-conditioning
All-Cause Mortality (participants affected / at risk) | 10/45 | 5/30
Serious Adverse Events (participants affected / at risk) | 28/45 | 20/30
Other Adverse Events (participants affected / at risk) | 41/45 | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-conditioning (N=45) | Post-conditioning (N=30)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Eye movement disorders (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Condition aggravated (General disorders) | 7 | 2
Multiple organ dysfunction (General disorders) | 4 | 2
Pyrexia (General disorders) | 1 | 3
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Acute GVHD in intestine (Immune system disorders) | 0 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 0
Engraftment syndrome (Immune system disorders) | 0 | 2
Septic shock (Infections and infestations) | 4 | 3
Pneumonia (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Enterococcal sepsis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Gianotti-Crosti syndrome (Infections and infestations) | 1 | 0
Histoplasmosis disseminated (Infections and infestations) | 1 | 0
Necrotizing fasciitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
BSCT failure (Injury, poisoning and procedural complications) | 0 | 1
Engraft failure (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Cerebral disorders (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Subdural hygroma (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-conditioning (N=45) | Post-conditioning (N=30)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 3 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 4
Bradycardia (Cardiac disorders) | 4 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 8 | 3
Abdominal distension (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 6
Nausea (Gastrointestinal disorders) | 0 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 6
Vomiting (Gastrointestinal disorders) | 5 | 6
Asthenia (General disorders) | 3 | 0
Condition aggravated (General disorders) | 18 | 1
Mucosal inflammation (General disorders) | 1 | 8
Oedema (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 3 | 0
Pain (General disorders) | 6 | 3
Pyrexia (General disorders) | 14 | 15
Graft versus host disease (Immune system disorders) | 0 | 2
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 2
Graft versus host disease in liver (Immune system disorders) | 0 | 2
Graft versus host disease in skin (Immune system disorders) | 0 | 5
BK virus infection (Infections and infestations) | 0 | 2
Clostridium difficile infection (Infections and infestations) | 3 | 1
Cytomegalovirus infection (Infections and infestations) | 4 | 5
Otitis externa (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 3 | 0
Adenovirus test positive (Investigations) | 0 | 2
Blood immunoglobulin G decreased (Investigations) | 1 | 2
Human rhinovirus test positive (Investigations) | 0 | 3
Polyomavirus test positive (Investigations) | 0 | 2
Transaminases increased (Investigations) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 4
Hypomagnesaemia (Investigations) | 3 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Agitation (Psychiatric disorders) | 2 | 2
Irritability (Psychiatric disorders) | 5 | 3
Renal failure (Renal and urinary disorders) | 0 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 7 | 6
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 2
Hypertension (Vascular disorders) | 19 | 9
Hypotension (Vascular disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: US protocol (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT01818492/Prot_000.pdf
  • Study Protocol: EU protocol (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT01818492/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT01818492/SAP_002.pdf